CLINICAL TRIAL: NCT03015337
Title: Relationship of Motor Skill Competency and Physical Fitness to Physical Activity in Elementary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Associate professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HUM00088758
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- New Physical Education Instructions (Experimental)
  Interventions: Behavioral: New physical education instructions

INTERVENTIONS:
Behavioral: New physical education instructions

SUMMARY:
This study examined how well elementary students demonstrated motor skill competency as a result of participating in the evidence-based quality physical education program and investigated relationships between levels of health-related physical fitness and physical activity in school-aged children.

ELIGIBILITY:
Inclusion Criteria:

* K-5 th grade students who are enrolled in 9 elementary schools in Southeast Michigan.

Exclusion Criteria:

-

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1844 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Running skill assessment | 2 years
  changes in manipulative skill between the intervention year 1 and the intervention year 2. The K-1 students' motor skill competency in running, weight transferring, hand dribbling, and underhand catching skills was assessed using four PE Metrics skill assessment rubrics in the intervention year 1 and year 2, respectively.
Weight transferring skill assessment | 2 years
  changes in manipulative skill between the intervention year 1 and the intervention year 2. The K-1 students' motor skill competency in running, weight transferring, hand dribbling, and underhand catching skills was assessed using four PE Metrics skill assessment rubrics in the intervention year 1 and year 2, respectively.
hand dribbling skill assessment | 2 years
  changes in manipulative skill between the intervention year 1 and the intervention year 2. The K-1 students' motor skill competency in running, weight transferring, hand dribbling, and underhand catching skills was assessed using four PE Metrics skill assessment rubrics in the intervention year 1 and year 2, respectively.
underhand catching skill assessment | 2 years
  changes in manipulative skill between the intervention year 1 and the intervention year 2. The K-1 students' motor skill competency in running, weight transferring, hand dribbling, and underhand catching skills was assessed using four PE Metrics skill assessment rubrics in the intervention year 1 and year 2, respectively.
FitnessGram test | 1 year
  Relationship between fitness and physical activity.
Daily physical activity participation in minutes | 1 year
  Relationship between levels of fitness and daily physical activity participation.

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Chen, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- School of Kinesiology, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen W, Hammond-Bennett A, Hypnar A, Mason S. Health-related physical fitness and physical activity in elementary school students. BMC Public Health. 2018 Jan 30;18(1):195. doi: 10.1186/s12889-018-5107-4. PMID 29378563
- [Derived] Chen W, Hammond-Bennett A, Hypnar A. Examination of motor skill competency in students: evidence-based physical education curriculum. BMC Public Health. 2017 Feb 23;17(1):222. doi: 10.1186/s12889-017-4105-2. PMID 28228116